CLINICAL TRIAL: NCT07169903
Title: Comparison of Segmentectomy Versus Lobectomy for Lung Adenocarcinoma 2 - 3cm With IASLC Grade 1 - 2 by Intraoperative Frozen Sections: A Prospective and Multi - Center Randomized Controlled Trial Study
Brief Title: Segmentectomy vs Lobectomy for 2 - 3cm IASLC Grade 1-2 Lung Adenocarcinoma: A Multi-center RCT
Acronym: STAR012
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Affiliated Hospital of Nantong University (Other); Huadong Hospital (Other); Anhui Chest Hospital (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); Center hospital of Nanyang (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Huzhou Central Hospital (Other); Anhui Provincial Hospital (Other Government); Shandong Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Chang Chen, Professor at Tongji University School of Medicine and Chief Physician of the Department of Thoracic Surgery at Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR012
Record Dates: First submitted 2025-06-15; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Lung Adenocarcinoma
Keywords: Segmentectomy; Lobectomy; Lung Adenocarcinoma; IASLC Grade; Randomized Controlled Trial
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lobectomy Group (No Intervention): Lobectomy includes resection of the right upper or lower lobe, and the left upper or lower lobe. Resection of more than one pulmonary lobe does not meet the criteria. The surgical margin, that is, the distance between the cut end covered by the visceral pleura and the tumor edge, is evaluated macroscopically to confirm that the surgical margin is not less than the maximum diameter of the tumor or 20 mm. If there is no frozen pathological diagnosis or cytological examination, it is necessary to confirm that there is no tumor residue at the margin before closing the chest. If the resection margin is positive for residual tumor cells, further surgical resection beyond the planned procedure must be performed.
- Segmentectomy group (Experimental): Segmentectomy involves resection of a pulmonary segment or a segment along with its adjacent segments. After segmentectomy, the surgical margin is examined macroscopically by evaluating the distance between the cut end covered by the visceral pleura and the tumor edge. If the surgical margin is smaller than the maximum diameter of the tumor or 20 mm, or if the margin is positive for residual tumor cells, the resection scope should be expanded. If the margin remains positive after expansion, segmentectomy should be converted to lobectomy.
  Interventions: Procedure: Pulmonary segmentectomy

INTERVENTIONS:
Procedure: Pulmonary segmentectomy — Segmentectomy is applied to lung adenocarcinomas with a diameter of 2-3 cm, in which intraoperative frozen pathology confirms a new pathological grade of 1-2.
  Other Names: Segmentectomy
  Arms: Segmentectomy group

SUMMARY:
This study is a prospective, multicenter randomized controlled trial (RCT) designed to compare the efficacy of segmentectomy and lobectomy for invasive lung adenocarcinoma with a diameter of 2-3 cm and intraoperative frozen section-confirmed IASLC pathological new grade 1-2. The non-inferiority of segmentectomy is primarily evaluated by 5-year relapse-free survival (RFS) and overall survival (OS) after surgery, while secondary endpoints include pulmonary function preservation, perioperative complications, etc. With a planned enrollment of 587 patients over a 3-year recruitment period and a 5-year follow-up, this study aims to identify an optimized surgical approach.

DETAILED DESCRIPTION:
Lung cancer is the most prevalent and lethal malignant tumor worldwide. Surgical resection remains the most effective treatment for early-stage lung cancer, with lobectomy historically serving as the standard procedure. Recent studies have demonstrated that segmentectomy can achieve comparable outcomes to lobectomy for tumors ≤2 cm and those with ground-glass opacity dominance (CTR ≤0.5). However, for invasive lung adenocarcinomas measuring 2-3 cm with solid predominance (CTR >0.5), high-level evidence supporting segmentectomy as an alternative to lobectomy is lacking. The 2020 International Association for the Study of Lung Cancer (IASLC) proposed a new grading system for invasive adenocarcinoma, which stratifies prognosis based on histologic subtypes. Tumors with IASLC Grade 1-2 (≤20% high-grade components) have better outcomes, but their optimal surgical approach (segmentectomy vs. lobectomy) in solid-predominant lesions (2-3 cm) remains unproven. Intraoperative frozen section has shown high accuracy in diagnosing IASLC grades, enabling real-time surgical decision-making. The primary objective of this study is to evaluate whether segmentectomy is non-inferior to lobectomy in terms of 5-year relapse-free survival (RFS) and overall survival (OS) for patients with 2-3 cm lung adenocarcinomas confirmed as IASLC Grade 1-2 by intraoperative frozen section.

ELIGIBILITY:
1. Initial Registration (1.1) Inclusion Criteria: 1. Aged 20 to 79 years, regardless of gender. 2. Preoperative CT or PET-CT suggests: ① Imaging diameter of 2-3 cm.

   * Suspicion of non-small cell lung cancer (NSCLC).

     * Solitary nodule or concomitant lesions with microinvasion or below.

       * Primary tumor not located in the middle lobe.

         * No suspected lymph node involvement. 3. Preoperative CT lung window (window level -700HU, window width 1500HU) indicates the nodule is predominantly solid, i.e., the consolidation-to-tumor ratio (CTR) is greater than 0.5 (CTR > 0.5).

           4. Good lung function (FEV1 > 1.5 L or FEV1% ≥ 60%), tolerable for both segmentectomy and lobectomy.

           5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. 6. Voluntary participation with signed informed consent, able to comply with study visit plans and other protocol requirements.

           7. No history of ipsilateral thoracotomy; video-thoracoscopic examination meets the criteria.

           8. No history of chemotherapy or radiotherapy, including treatment for other cancers. Eligible if more than 5 years have passed since completion of perioperative adjuvant chemotherapy. Eligible if there is a history of or ongoing hormone therapy.

           9. All the following laboratory test results are eligible (all laboratory tests use the latest results within 28 days before initial registration; laboratory tests on the same day within 4 weeks before initial registration are allowed):
           * White blood cell count ≥ 3000/mm³.
   * Hemoglobin ≥ 8.0 g/dL (without blood transfusion within 28 days before initial registration).

     * Platelet count ≥ 10×10⁴/mm³.

       * AST ≤ 100 IU/L.

         ⑤ ALT ≤ 100 IU/L.

         ⑥ Total bilirubin ≤ 2.0 mg/dL.

         ⑦ Serum creatinine ≤ 1.5 mg/dL. 10. The patient has signed a written informed consent. (1.2) Exclusion Criteria:
         1. Active bacterial or fungal infection (confirmed by imaging diagnosis or bacteriological examination with fever >38°C).
         2. Multiple active cancers (synchronous or metachronous multiple primary cancers, excluding in situ carcinoma or intramucosal cancer lesions considered cured by local treatment; such lesions are not included in active multiple cancers).
         3. Patients with severe impairment of cardiac, hepatic, or renal function (cardiac function grade 3-4; ALT and/or AST more than 3 times the upper limit of normal; Cr exceeding the upper limit of normal).
         4. Patients with concomitant other malignant tumors or hematological diseases.
         5. Pregnant, planning to become pregnant, or lactating female patients (diagnosed with early pregnancy when urine HCG >2500 IU/L).
         6. Any form of antitumor therapy before tumor resection, including interventional chemotherapy embolization, ablation, radiotherapy, chemotherapy, and molecular targeted therapy.
         7. Patients who participated in other tumor-related clinical trials within the past three months.
         8. Preoperative CT suggests ground-glass predominant nodules (CTR < 0.5).
         9. Patients with positive lymph nodes indicated by preoperative imaging or lymph node puncture (clinical N stage = 1 or 2).
         10. Patients with tumors near the hilum who cannot undergo segmentectomy.
         11. Patients deemed unsuitable for enrollment by the investigator.
2. Intraoperative Secondary Registration (2.1) Inclusion Criteria: 1. Intraoperative frozen section indicates invasive lung adenocarcinoma with International Association for the Study of Lung Cancer (IASLC) grade 1-2 (<20% pathological high-grade subtypes).

2. Intraoperative frozen section shows negative surgical margins. 3. Intraoperative exploration reveals no severe adhesions or lymph node inflammatory changes (adhesions of pulmonary vessels or bronchi), confirming feasibility for both lobectomy and segmentectomy.

(2.2) Exclusion Criteria:

1. Patients with IASLC grade 3 (≥20% pathological high-grade subtypes) indicated by intraoperative frozen section.
2. Patients confirmed with in situ carcinoma or microinvasive adenocarcinoma by intraoperative frozen section.
3. Patients with preoperative findings of distant metastasis or pleural/ascitic effusion.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Overall Survival (OS) is defined as the time from the date of surgery to death from any cause. For surviving patients, survival time is censored at the last date when survival was confirmed; the study allows telephone confirmation of survival status, provided that medical records are available. For lost-to-follow-up patients, survival time is censored on the last date when survival was confirmed before the loss of follow-up. For patients diagnosed with non-malignant tumors, the date of surgery is used as the censorship point.
Recurrence-Free Survival (RFS) | 5 years
  Recurrence-Free Survi refers to the time from the date of surgery to the diagnosis of recurrence or death from any cause, whichever occurs first. "Recurrence" includes both cases confirmed by imaging diagnosis and clinical exacerbation (symptomatic aggravation) not confirmed by imaging diagnosis. For the former, the day of imaging examination is regarded as the recurrence date, while for the latter, the day of diagnosing symptomatic deterioration is considered the recurrence date. An increase in tumor marker values alone is not considered an RFS event. When recurrence is confirmed based on the pathological results of a biopsy specimen, if the patient had already been clinically diagnosed with recurrence before, the endpoint is the date of clinical diagnosis; otherwise, it is the biopsy date. The occurrence of other primary cancers is not considered an endpoint, and RFS continues until other events are identified.

SECONDARY OUTCOMES:
Postoperative Respiratory Function | 12 months
  Patients underwent respiratory function tests (forced expiratory volume in 1 second) at 6 months and 12 months postoperatively to assess the differences between baseline respiratory function and that at 6 months and 12 months postoperatively.
Hospitalization Duration | 1 month
  The hospitalization duration was calculated as the median number of days from the date of surgery.
Chest Tube Placement Time | 1 month
  The chest tube placement time is calculated as the median number of days from the surgery date to chest tube removal. If the chest tube is placed after the patient's discharge, the placement time is calculated until the tube is removed. If the patient undergoes a second chest tube placement, the time after replacement is not included in the calculation.
Surgical Time | 1 day
  The surgical time is calculated as the duration from incision to the end of the operation.
Blood Loss | 1 day
  The blood loss is measured from the incision to the end of the operation and recorded in milliliters (mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No